CLINICAL TRIAL: NCT05733546
Title: A Phase II, Multicentre, Randomised, Double-blind, Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of COMP360 in Participants With Recurrent Major Depressive Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: COMPASS Pathways (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMP 104
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: psilocybin, MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 25 mg COMP360 Psilocybin (Experimental): 25 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin
- 10 mg COMP360 Psilocybin (Experimental): 10 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin
- 1 mg COMP360 Psilocybin (Active Comparator): 1 mg COMP360 Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — COMP360 Psilocybin administered under supportive conditions
  Other Names: COMP360

SUMMARY:
Safety, Tolerability, pharmacokinetics and efficacy of a single administration of COMP360 in participants with recurrent Major Depressive Disorder.

DETAILED DESCRIPTION:
This is a phase II, multi-centre, randomised, double-blind, controlled study. The study population will include participants aged ≥18 years with recurrent Major Depressive Disorder (MDD) with up to four prior treatment failures of an antidepressant in their current depressive episode.

Overall, 102 participants will be randomised in a 1:1:1 ratio to receive COMP360 25 mg, COMP360 10mg or COMP360 1 mg.

In this study the aim is to investigate the safety and tolerability of COMP360, administered with psychological support, in adult participants with MDD with one prior treatment failure. In addition, pharmacokinetics and efficacy of COMP360 will be investigated.

The study will last up to 16 weeks including a three- to ten-week Screening Period and a six-week follow-up from investigational product (IP) administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged ≥18 years at Screening
* Major depression without psychotic features (single or recurrent episode as informed by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition [DSM-5])
* If the current major depressive episode is the participant's first lifetime episode of depression, the length of the current episode must be ≥3 months and ≤2 years at Screening
* MADRS total score ≥20 at Screening and Baseline to ensure at least moderate severity of depression.
* Failure to respond to an adequate dose and duration of up to four pharmacological treatment for the current episode as determined through the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and using the supplementary advice on additional antidepressants not included in MGH-ATRQ.
* At Screening, agreement to discontinue all prohibited medications.

Key Exclusion Criteria:

* Prior or ongoing bipolar disorder, any psychotic disorder, including schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder (unless substance induced or due to a medical condition), antisocial personality disorder as assessed by a structured clinical interview (MINI 7.0.2)
* Lifetime paranoid, schizoid, schizotypal, histrionic, narcissistic personality disorder, or any ongoing serious psychiatric comorbidity based on medical history and clinical judgement
* Borderline personality disorder as demonstrated by medical history or the Mini International Neuropsychiatric Interview Plus (MINI plus) - borderline personality disorder module
* Ongoing post-traumatic stress disorder, obsessive-compulsive disorder, or anorexia nervosa as assessed by medical history and a structured clinical interview (MINI 7.0.2) Psychiatric inpatient within the past 12 months prior to Screening
* Use of electroconvulsive therapy, deep brain stimulation, or vagus nerve stimulation during the current depressive episode
* Transcranial magnetic stimulation within the past six months prior to Screening
* Current enrolment in a psychological therapy programme that will not remain stable for the duration of the study. Psychological therapies cannot have been initiated within 30 days prior to Screening
* Exposure to COMP360 psilocybin therapy prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of COMP360 Psilocybin | Up to Week 6
  Proportion of patients with adverse events (AEs)

SECONDARY OUTCOMES:
Pharmacokinetics of COMP360 Psilocybin | Day 1
  Plasma concentrations of psilocybin, psilocin, 4-hydroxyindoleacetic acid (4-HIAA) and psilocin-O-glucuronide post-COMP360 administration on Day 1
Change from baseline in MADRS total score at Week 3 and Week 6 for COMP360 25 mg versus COMP360 1 mg | Week 3 and Week 6
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Kadima Neuropsychiatry Institute, La Jolla, California
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Sunstone Therapies, Rockville, Maryland
  - Elixia MA, LLC, Springfield, Massachusetts
  - Aims Trial, Plano, Texas

IPD SHARING:
Plan to Share IPD: No